CLINICAL TRIAL: NCT07036107
Title: Robotic-SNS: A Multicenter, Randomized Trial on the Clinical and Socioeconomic Impact of Wearable Exoskeletons for Spinal Cord Injury Rehabilitation in the Spanish Healthcare System
Brief Title: A Trial on the Clinical and Socioeconomic Impact of Wearable Exoskeletons for Spinal Cord Injury Rehabilitation in the Spanish Healthcare System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ABLE Human Motion S.L. (Industry)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other); Universitat de Lleida (Other); Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Robotic-SNS
Record Dates: First submitted 2025-06-06; First posted 2025-06-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic exoskeleton (Experimental): The intervention group will receive rehabilitation treatment with the ABLE Exoskeleton
  Interventions: Device: ABLE Exoskeleton
- Conventional therapy (Active Comparator): The control group will receive conventional therapy for gait rehabilitation
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: ABLE Exoskeleton — Participants will receive a 24-session rehabilitation treatment program with the ABLE Exoskeleton, 3 times a week for up to 8 weeks
  Arms: Robotic exoskeleton
Other: Conventional therapy — Participants will receive a 24-session conventional therapy program for gait rehabilitation, 3 times a week for up to 8 weeks.
  Conventional therapy includes joint mobilizations, strengthening of paretic muscles and re-education of walking with parallel bars, making use of the technical aids and orthoses required by the patient (KAFOs, crutches and walkers).
  Arms: Conventional therapy

SUMMARY:
This clinical trial aims to collect evidence on the clinical benefits and the socioeconomic impact of integrating a novel wearable powered lower-limb exoskeleton for gait rehabilitation in acute/subacute spinal cord injured individuals and to evaluate the efficiency of this technology to the current standard of care in the Spanish Healthcare System (SNS).. The main questions it aims to answer are:

* Is robotic therapy for gait rehabilitation more effective and efficient than conventional therapy?
* Does robotic therapy for gait rehabilitation reduce the burden on healthcare professionals and caregivers?
* Does robotic therapy for gait rehabilitation reduce direct healthcare costs?
* Does robotic therapy for gait rehabilitation reduce intervention-related costs?

Researchers will compare a novel wearable powered lower-limb exoskeleton for gait rehabilitation to conventional therapy to see if the robotic exoskeleton is more effective and efficient in improving clinical benefits and to assess if it reduces the burden of healthcare professionals and caregivers, as well as healthcare and intervention-related costs.

Participants will:

* Be randomized on a 1:1 basis to receive rehabilitation treatment with either the robotic exoskeleton or conventional therapy for gait recovery, 3 times a week on non-consecutive days for 8 weeks (24-session program).
* Undergo a pre- and post-intervention assessment of clinical, functional, physiological, psychological, and socioeconomic variables.
* Have a follow-up visit 2 months after the end of the treatment.

DETAILED DESCRIPTION:
Participants will be recruited from among patients admitted to the institutions involved in the project: Vall d'Hebron University Hospital (HVH) through its research institute (VHIR) and the National Hospital for Paraplegics of Toledo (HNP), through its research foundation (FHNP). After checking the inclusion and exclusion criteria, informing the patient and signing the consent, they will be randomly distributed between the control group (CG) and the intervention group (IG). Open random parallel groups. The IG will receive rehabilitation treatment with the ABLE Exoskeleton, while the CG will receive conventional therapy for gait rehabilitation. The latter includes joint mobilizations, strengthening of paretic muscles and re-education of walking with parallel bars, making use of the technical aids and orthoses required by the patient (KAFOs, crutches and walkers). For both groups, participation in the study is based on a baseline visit, the 24-session rehabilitation treatment (including mid-training and end-training assessments at 12-session and 24-session, respectively) and a follow-up visit two months after the end of the treatment. Caregiver overload will also be assessed at baseline visit, after patient's treatment and at the follow-up visit two months after patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of spinal cord injury (SCI) in the acute or subacute phase (< 6 months of evolution)
* traumatic or non-traumatic aetiology
* neurological level of the SCI between C5 and L5 for patients with American Spinal Injury Association Impairment Scale (AIS) C or D, and SCI between C7 and L5 for patients with AIS A or B.
* sufficient strength in the upper extremities to handle a walker (triceps muscle score ≥ 4 according to the Medical Research Council (MRC) scale).
* range of motion (ROM) without limitations in the lower extremities (achieve at least a knee extension of 10 degrees and neutral ankle position)
* muscle spasticity in the lower extremities with a score ≤ 3 on the Modified Ashworth Scale (MAS)
* tolerate bipedalism (having stood up in the last year)
* aged between 18 and 70 years, with height between 150 cm and 190 cm, and weight less than 100 kg

Exclusion Criteria:

* WISCI ≥ 15
* cognitive or neurological limitations that prevent following instructions
* another neurologic disorder permanently affecting gait and gait therapy (other than SCI)
* grade I or higher in the European Pressure Ulcer Advisory Panel (EPUAP) in the areas of contact with the exoskeleton
* unresolved fractures at the time of the study
* uncontrolled autonomic dysautonomia
* intolerance to exercise
* uncontrolled epilepsy
* previous experience with Robotic-Assisted Gait Training (RAGT).
* ROM restriction such as flexing or arthrodesis will be excluded
* spinal instability (or spinal orthotics unless cleared by a medical doctor).
* deterioration >3 points of the total in the motor score of the International Standards for the Neurological Classification of Spinal Cord Injury (ISNCSCI) in the last 4 weeks. Loss of sensation and/or motor activity above the level of injury detected that has not been evaluated by a doctor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Walking ability | Baseline , end of treatment (at 8 weeks), and follow-up (2 months after end of treatment)
  The walking ability will be assessed using the Walking Index Spinal Cord Injury (WISCI) II which evaluates the amount of physical assistance needed, as well as devices required, for walking following paralysis that results from Spinal Cord Injury (SCI).
  The WISCI II score ranges from 0 to 20 (0: the individual is unable to walk, 20: the individual walks without assistance or devices)
Change in Balance | Baseline, mid-training (at 4 weeks), and end of treatment (at 8 weeks)
  The balance will be assessed by the time taken to complete the Timed-Up-and-Go (TUG) test which evaluates mobility and balance.
Change in Gait speed | Baseline, mid-training (at 4 weeks), and end of treatment (at 8 weeks)
  The gait speed will be assessed by the time taken to complete the 10 meter Walk Test (10mWT) which evaluates walking speed in meters per second over a short duration.
Change in Lower Extremity Motor Score (LEMS) | Baseline, mid-training (at 4 weeks), end of treatment (at 8 weeks), and follow-up (2 months after end of treatment)
  The Lower Extremity Motor Score (LEMS) evaluates motor function on a scale of 0 (no motor function) to 5 (full motor function) for 5 lower extremity muscle groups with a 50-point maximum (25 per side).
Change in Trunk control | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after end of treatment)
  The trunk control will be assessed using the Trunk Assessment Scale for Spinal Cord Injury (TASS). The TASS consists of nine sitting tasks without upper-limb support: one task is static, and the other eight tasks are dynamic. Each item is assigned a score of 0-2, 0-4, or 0-6 for a total score of 44, with higher scores indicating better trunk function.
Change in Endurance | Baseline, mid-training (at 4 weeks), and end of treatment (at 8 weeks)
  Endurance will be assessed by the distance (in meters) walked during the 2-Minute Walk Test (2MWT), which evaluates walking capacity and functional mobility.
Change in Endurance | Baseline, mid-training (at 4 weeks), and end of treatment (at 8 weeks)
  Endurance will be assessed by the distance (in meters) walked during the 6-Minute Walk Test (6MWT), which evaluates walking capacity and functional mobility.
Change in Level of Exertion | Baseline, mid-training (at 4 weeks), and end of treatment (at 8 weeks)
  Perceived exertion associated with the walking test (2MWT/6MWT) will be assessed using the Borg Rating of Perceived Exertion Scale, a self-report scale ranging from 0 to 10. A score of 0 indicates no exertion, and 10 indicates maximal exertion. Higher scores represent greater perceived exertion.
Change in Gait pattern | Baseline, mid-training (at 4 weeks), end of treatment (at 8 weeks), and follow-up (2 months after end of treatment)
  The gait pattern and compensatory movements will be assessed through kinetic and kinematic gait parameters collected using a 3-D gait analysis system. The Gait Deviation Index for SCI (SCI-GDI) will be calculated to evaluate the difference between the patient' gait pattern compared to the reference gait pattern.
  The SCI-GDI score typically ranges from 0 to 100, with 100 representing a normal gait pattern.
Change in Bladder and Bowel function | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after end of treatment)
  Bladder and bowel function will be assessed using the International Standards to document Autonomic Function following SCI (ISAFSCI), which identifies which autonomic functions (e.g., bladder, bowel) are intact, impaired, or lost.
Change in Bladder and Bowel function | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after end of treatment)
  Bowel function will also be assessed using the Neurogenic Bowel Dysfunction score (NBD score), a self-report questionnaire.
  The total NBD score ranges from 0 to 47, with higher scores indicating more severe dysfunction.
Change in Bone density | At baseline and end of treatment (at 8 weeks)
  The Bone density will be assessed through analytical control, 24-hour urine, and dual-energy X-ray absorptiometry (DEXA) scan in the spine, hip and knee.
Change in Cardiovascular function | At baseline and end of treatment (at 8 weeks)
  The cardiovascular function will be asssessed by an arm ergometry test, which is a test that measures the heart's response to physical exertion. The maximum heart rate (HR) will be documented.
Change in Respiratory function | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after end of treatment)
  The respiratory function will be assessed by a simple spirometry, which is a test that measures the volume of air exhaled in one second (FEV1) and the total volume of air exhaled forcefully (FVC).
Pain reduction | From baseline to follow-up (at 2 months after the end of treatment)
  The reduction in pain will be assessed using International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) which is used to document the interference of pain with physical and emotional function and sleep, probable pain diagnosis, location, intensity and duration.
  Each value is scored on a 0 to 10 numerical rating scale, where 0 represents no pain and 10 represents the worst pain imaginable.
Change in Spasticity | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after the end of treatment)
  The spasticity in the lower limbs will be assessed using both the Spinal Cord Assessment Tool for Spastic Reflexes (SCATS) score, which evaluates three types of spastic motor behaviors in SCI patients - clonus, flexor spasms, and extensor spasms, as well as the Modified Ashworth Scale (MAS).
  SCATS total score (0-9; higher = worse outcome)
Change in Functional independence | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after the end of treatment)
  The functional independence will be assesed using the Spinal Cord Independence Measure III (SCIM III) which is a patient-reported outcome measure that evaluates three main domains: self-care, respiration and sphincter management, and mobility. The SCIM III score is calculated on a scale of 0-100, with 0 indicating complete dependence and 100 indicating complete independence.
Change in Quality of Life | At baseline and end of treatment (at 8 weeks)
  Quality of life will be assessed using the 5-level EQ-5D version (EQ-5D-5L), a standardized instrument for measuring generic health status.
  Ranging from 1 (best possible health) to values less than 0.
Change in Quality of Life | At baseline and end of treatment (at 8 weeks)
  Emotional well-being will be assessed using the Hospital Anxiety and Depression Scale (HADS), which measures anxiety and depression.
  Score on HADS subscales (0-21 per subscale; with higher numbers indicating a greater level of anxiety or depression)
Change in Quality of Life | At baseline and end of treatment (at 8 weeks)
  Motivation will be assessed using the interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMI).
  Interest/Enjoyment score on IMI subscale (1-7; where 1 represents "Not at all true" and 7 represents "Very true")
Burden of healthcare professionals | At end of treatment (8 weeks)
  The burden on healthcare professionals will be assessed using the NASA Task Load Index (NASA-TLX), a self-report questionnaire to assess work load on five 7-point scales. NASA-TLX scores can range from 0 to 100, where a higher score generally indicates a higher workload
Change in Burden of the caregiver | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after the end of treatment)
  The caregiver burden will be assessed using the Zarit Burden Interview, a 22-item self-report questionnaire which total score ranges from 0 to 88. The higher the value, the higher the caregiver burden.
Change in Direct healthcare costs | Baseline (Day 0), end of treatment (8 weeks), and follow-up (16 weeks)
  The medical costs including hospitalization days, transportations, specialists consultations, rehabilitation services, emergency room visits, and hospital admissions will be calculated.
Intervention-related costs | At the end of treatment (8 weeks)
  The costs associated to the rehabilitation sessions, treatment, and equipment during the intervention period will be calculated.
Change in the productivity losses | Baseline, end of treatment (at 8 weeks), and follow-up (2 months after the end of treatment)
  Variation in indirect costs for patient and caregiver, associated with reduced work capacity, absenteeism, or early retirement, as a result of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lluïsa Montesinos Magraner, Dr, Principal Investigator — Hospital Universitario de Vall d'Hebron; Ana de los Reyes Guzmán, PhD, Principal Investigator — Hospital Nacional de Parapléjicos
Locations (2):
- Spain (2):
  - Hospital Nacional de Parapléjicos, Toledo, Castille-La Mancha
  - Hospital Universitario de Vall d'Hebron, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No